CLINICAL TRIAL: NCT00524251
Title: The Effect of Lifestyle-Adjustments Prior to Medical Treatment on the Effect of Medical Treatment in Reflux Patients
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Other Study IDs: N11
Record Dates: First submitted 2007-08-29; First posted 2007-09-03 (Estimated); Last update posted 2008-09-17 (Estimated); Status verified 2008-09

CONDITIONS: GERD; Quality of Life
Keywords: Patients with reflux complaints; GERD; quality of life; lifestyle adjustments
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Esomeprazole

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: esomeprazole

SUMMARY:
The purpose of this study is to determine whether the improvement in the quality of life after an initial treatment with esomeprazole 40mg for reflux disease is the same in patients who have already made lifestyle-adjustments as in patients who have not implemented lifestyle-adjustments prior to the start of treatment (baseline)

ELIGIBILITY:
Inclusion Criteria:

* Patients with reflux complaints
* 18 years of age

Exclusion Criteria:

* Restrictions as mentioned in the registration text
* H2RA or PPI use in the month prior to inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 990 (Estimated)
Dates: Start 2004-06; Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: A Sellink, MD, Study Director — AstraZeneca; N van den Berk, Study Chair — AstraZeneca
Locations (54):
- Netherlands (54):
  - Research Site, 's-Gravenzande
  - Research Site, Almere Stad
  - Research Site, Apeldoorn
  - Research Site, Baarn
  - Research Site, Bennebroek
  - Research Site, Blaardingen
  - Research Site, Boekel
  - Research Site, Delft
  - Research Site, Enschede
  - Research Site, Ewijk
  - Research Site, Geleen
  - Research Site, Haelen
  - Research Site, Halfweg NH
  - Research Site, Hardenberg
  - Research Site, Heemstede
  - Research Site, Hillegom
  - Research Site, Hilversum
  - Research Site, Horst
  - Research Site, Kerkrade
  - Research Site, Klimmen
  - Research Site, Landgraaf
  - Research Site, Laren
  - Research Site, Leusden
  - Research Site, Lichtenvoorde
  - Research Site, Lisse
  - Research Site, Maastricht
  - Research Site, Monster
  - Research Site, Nieuw-Vennep
  - Research Site, Nieuwegein
  - Research Site, Nijverdal
  - Research Site, Ochten
  - Research Site, Oisterwijk
  - Research Site, Oldenzaal
  - Research Site, Pijnacker
  - Research Site, Rijnsburg
  - Research Site, Rijssen
  - Research Site, Schijndel
  - Research Site, Sittard
  - Research Site, Soest
  - Research Site, Spakenburg
  - Research Site, Susteren
  - Research Site, Swalmen
  - Research Site, The Hague
  - Research Site, Tilburg
  - Research Site, Vaals
  - Research Site, Valkenburg
  - Research Site, Veenendaall
  - Research Site, Velp
  - Research Site, Warnsveld
  - Research Site, Wassenaar
  - Research Site, Westerhaar-Vrienzenv Wijk
  - Research Site, Zandvoort
  - Research Site, Zevenhuizen
  - Research Site, Zoetermeer